CLINICAL TRIAL: NCT02658643
Title: Randomized Controlled Study to Determine the Difference in Time and Complication Rate for Biliodigestive Anastomosis by Continuous Versus Interrupted Suture Technique
Brief Title: Analysis of Biliodigestive Anastomosis Techniques (BDA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VTG-06
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Continuous or Interrupted Suture
Keywords: biliodigestive anastomosis techniques

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous suture technique (Experimental): The BDA is performed as continuous suture with two separate all-layer suture for the behind - and front-wall of the anastomosis
  Interventions: Procedure: Continuous suture technique
- Interrupted suture technique (Active Comparator): The BDA is performed as interrupted suture with two separate all-layer suture for the behind - and front-wall of the anastomosis
  Interventions: Procedure: Interrupted suture technique

INTERVENTIONS:
Procedure: Continuous suture technique — The BDA is performed as continuous suture with two separate all-layer suture for the behind - and front-wall of the anastomosis
  Arms: Continuous suture technique
Procedure: Interrupted suture technique — The BDA is performed as interrupted suture with two separate all-layer suture for the behind - and front-wall of the anastomosis
  Arms: Interrupted suture technique

SUMMARY:
The aim of this prospective randomized controlled study is to determine the benefit-risk ratio (success rate, complication rate, tolerance) for patients with biliodigestive anastomosis by either continuous or interrupted suture.

DETAILED DESCRIPTION:
The aim of this prospective randomized controlled study is to determine the benefit-risk ratio (success rate, complication rate, tolerance) for patients with biliodigestive anastomosis by either continuous or interrupted suture. A biliodigestive anastomosis is a surgical connection between the common bile duct (ductus choledochus) and the digestive tract to prevent interference of bile flow. Indications for a biliodigestive anastomosis include total or partial resection of the pancreas and duodenum (PPPD, Whipple procedure) for pancreatic tumors, tumors of the biliary tract or duodenum, and biliary tract reconstructions during liver transplantation or advanced liver resections. Furthermore a biliodigestive anastomosis can be required to manage the injury of the biliary tract and infectious and traumatic structures of the biliary tract. Biliodigestive anastomoses can be performed by continuous or interrupted suture. The aim of this study is to determine the difference between continuous and interrupted suture for biliodigestive anastomoses, as advantages and disadvantages of each technique have not been determined. Only patients receiving their first biliodigestive anastomosis will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Scheduled for elective BDA procedure
* Primary BDA procedure
* Diameter of DHC > 7mm
* Written consent

Exclusion Criteria:

* Previous BDA procedure
* Impaired mental state or language problems
* Lacking compliance
* Emergency procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Time to complete the biliodigestive anastomosis | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Reißfelder, MD, Principal Investigator — christoph.reissfelder@uniklinikum-dresden.de
Locations (1):
- Department of Visceral, Thoracic and Vascular Surgery, University Hospital Carl Gustav Carus, TU Dresden, Germany, Dresden, Germany

REFERENCES:
- [Derived] Seifert L, von Renesse J, Seifert AM, Sturm D, Meisterfeld R, Rahbari NN, Kahlert C, Distler M, Weitz J, Reissfelder C. Interrupted versus continuous suture technique for biliary-enteric anastomosis: randomized clinical trial. BJS Open. 2023 Jan 6;7(1):zrac163. doi: 10.1093/bjsopen/zrac163. PMID 36723996